CLINICAL TRIAL: NCT02455843
Title: A Multicenter, Randomized, Open-label Phase III Trial of Microwave Plus Chemotherapy Versus Chemotherapy for Advanced NSCLC
Brief Title: Microwave Plus Chemotherapy Versus Chemotherapy for Advanced NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xin Ye, Chairman of Chinese Anti-Cancer Association Professional Committee of lung cancer minimally invasive therapy combined therapy branch, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongPH Jinan
Record Dates: First submitted 2015-05-16; First posted 2015-05-28 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: microwave ablation; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Patients were divided into two groups: The microwave ablation plus chemotherapy group and the chemotherapy group.The former will be treated with microwave, followed by chemotherapy.The latter will be treated with chemotherapy alone.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microwave plus chemotherapy (Experimental): In combination group, patients will be treated with microwave ablation in primary tumor sites followed by chemotherapy （For non-squamous cell lung cancer，patients will be treated with pemetrexed，500mg/m2, d1, ivdrip, or docetaxel,75mg/m2, d1, ivdrip or gemcitabine 1250mg/m2, d1 d8, ivdrip,or novelbine 25mg/m2 d1 d8, ivdrip, paclitaxel 175mg/m2 d1 ivdrip plus cisplatin 75mg/m2, d1 d2, ivdrip or carboplatin with an area under the curve of 5 d1 ivdrip. For squamous cell lung cancer，patients will be treated with docetaxel,75mg/m2, d1, ivdrip or gemcitabine 1250mg/m2, d1 d8, ivdrip plus cisplatin 75mg/m2, d1 d2, ivdrip or carboplatin with an area under the curve of 5 d1 ivdrip；repeated every 3 weeks and up to 6 cycles are administrated ）
  Interventions: Other: Microwave ablation
- chemotherapy (Placebo Comparator): In chemotherapy group,patients will be treated with chemotherapy alone（For non-squamous cell lung cancer，patients will be treated with pemetrexed，500mg/m2, d1, ivdrip plus cisplatin 75mg/m2, d1 d2, ivdrip or carboplatin with a area uder the curve of 5 d1 ivdrip. For squamous cell lung cancer，patients will be treated with docetaxel,75mg/m2, d1, ivdrip or gemcitabine 1250mg/m2, d1 d8, novelbine 25mg/m2 d1 d8, ivdrip, paclitaxel 175mg/m2 d1 ivdrip plus cisplatin 75mg/m2, d1 d2, ivdrip or carboplatin with an area under the curve of 5 d1 ivdrip；repeated every 3 weeks and up to 6 cycles are administrated ）
  Interventions: Other: Microwave ablation

INTERVENTIONS:
Other: Microwave ablation — Patients assigned to the combination group will be treated with microwave in the primary tumor site

SUMMARY:
This study is a multicenter, randomized, open-label Phase III trial that compares microwave plus chemotherapy versus chemotherapy in patients with advanced non-small cell lung cancer. The primary endpoint is progression free survival (PFS) and the key secondary endpoint is overall survival (OS). A total of 275 eligible patients will be randomized to receive either microwave ablation combinated with first-line platinum-based doublet chemotherapy（138） or first-line platinum-based doublet chemotherapy（137） in a 1:1 ratio until patients. The response of microwave ablation will be assessed by the expert consensus for thermal ablation of primary and metastatic lung tumors. Tumor response and progression will be assessed according to Response Evaluation Criteria in Solid Tumors（RECIST）1.1.

DETAILED DESCRIPTION:
Patients will be randomized to treated with microwave ablation and chemotherapy or treated with chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced stage NSCLC (stage IIIB or IV) which is confirmed by histology or cytology methods.
2. Measurable disease other than the primary tumors site according to RECIST1.1.
3. Eastern Cooperative Oncology Group (ECOG) score of 0-2
4. Adequate organ function, defined as all of the following:

   1. Left ventricular ejection fraction >50% or within institution normal values.
   2. Absolute neutrophil count (ANC)>1500/mm3.
   3. Platelet count >75,000/mm3
   4. Estimated creatinine clearance>45m1/min.
   5. Total bilirubin<1.5 times institutional ULN (Patients with Gilbert's Syndrome total bilirubin must be <4 times institutional ULN).
   6. Aspartate amino transferase (AST) or alanine amino transferase (ALT) < three times the institutional upper limit of normal (ULN) (if related to liver metastases<five times institutional ULN).
5. Age ≥ 18 years.
6. Written informed consent that is consistent with International Conference on Harmonization (ICH)-Good Clinical Practice（GCP） guidelines.

Exclusion Criteria:

1. Previous anti-cancer treatments including chemotherapy, radiation therapy or targeted therapy..
2. Active symptomatic brain metastases. Dexamethasone therapy will be allowed if administered as a stable dose for at least 4 weeks before randomization.
3. Any other current malignancy or malignancy diagnosed within the past five (5) years.
4. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association （NYHA） classification of 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to randomisation.
5. Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
6. Women of child-bearing potential and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to study entry.
7. Female patients of childbearing potential who are nursing or are pregnant.
8. Patients unable to comply with the protocol in the opinion of the investigator.
9. Active hepatitis B infection (defined as presence of Hepatitis B DNA), active hepatitis C infection (defined as presence of Hepatitis C RNA) and/or known HIV carrier.
10. Known or suspected active drug or alcohol abuse in the opinion of the investigator.
11. Major surgery within 4 weeks of starting study treatment. Use of any investigational drug within 4 weeks of randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to 12 months after the last patient randomized
  From the start of chemotherapy or ablation to the date of progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Kai x Zhang, M.D, Principal Investigator — Tengzhou Center of People's Hospital; Jing w Bi, M.D., Principal Investigator — Jinan Military General Hospital
Locations (14):
- China (14):
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Dezhou People's Hospital, Dezhou, Shandong
  - The Second People's Hospital of Dezhou, Dezhou, Shandong
  - Jinan Military General Hospital, Jinan, Shandong
  - Affliated Hospital of Shandong Academy of Medical Sciences, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Affliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng Cancer Hospital, Liaocheng, Shandong
  - The People's Hospital of Pingyi Country, Linyi, Shandong
  - Affliated Hospital of Taishan Medical University, Taian, Shandong
  - The People's Liberation Army 88 Hospital, Taian, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Tengzhou center of people's hospital, Zaozhuang, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wei Z, Ye X, Yang X, Huang G, Li W, Wang J, Han X. Microwave ablation plus chemotherapy improved progression-free survival of advanced non-small cell lung cancer compared to chemotherapy alone. Med Oncol. 2015 Feb;32(2):464. doi: 10.1007/s12032-014-0464-z. Epub 2015 Jan 9. PMID 25572816